CLINICAL TRIAL: NCT06710951
Title: Effect of Povidone-iodine 5% Vs 1% on the Ocular Surface As Antiseptic for Anti Vascular Endothelial Growth Factor Intravitreal Injections
Brief Title: Effect of Povidone-iodine 5% Vs 1% on the Ocular Surface in Intravitreal Injections of Anti-VEGF
Acronym: anti-VEGF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Gerardo García Aguirre (Other)
Responsible Party: Sponsor-Investigator, José Gerardo García Aguirre, Retina Adjunct, Asociación para Evitar la Ceguera en México
Organization: Asociación para Evitar la Ceguera en México (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RE-21-02
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye
Keywords: Povidone-iodine; Pain
MeSH Terms: conditions — Dry Eye Syndromes; Pain

STUDY DESIGN:
Intervention Model Description: Clinical, prospective, randomized trial. Pre anti-VEGF intravitreal injection, with OCULUS Keratopgrapph 5M topograph, non invasive tear breaking time, bulbar redness, and Oxford scale with fluorescein staining were measured. During anti-VEGF injection, tetracaíne was use as anestetic. Povidone-iodine 1% or 5% was randomized as antiseptic. After anti-VEGF intravitreal injection, patients were examined again for tear bkreaking time, bulbar redness and Oxford sacle, plus pain 15 minutes after injection. Finally, two days after the injection, patients were interviwed by telephone about their pain.
Who Masked: Participant
Masking Description: Patients did not know which percentage of povidone-iodine was utilized during their injection.
  Tear breaking time and bulbar redness were automized results by Keraatopgrah. Oxford scale pre and post injection was staged by an investigator that did not know the group in which the patient was.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone-iodine 1% (Experimental): Povidone-iodine 1% was used as antiseptic during anti-VEGF intravitreal injection
  Interventions: Procedure: Change of normal concentration of povidone-iodine 5% to 1%
- Povidone-iodine 5% (Active Comparator): Povidone-iodine 5% was used as antiseptic during anti-VEGF intravitreal injection
  Interventions: Procedure: Change of normal concentration of povidone-iodine 5% to 1%

INTERVENTIONS:
Procedure: Change of normal concentration of povidone-iodine 5% to 1% — Normal concentration of povidone-iodine during anti-VEGF intravitreal injection was 5%. That concentration was utilized in the control group, and 1% in the experimental group.

SUMMARY:
Objective and subjective comparison between the use of povidone-iodine 1% vs 5% as antiseptic in patients that need anti-VEGF intravitreal injection

DETAILED DESCRIPTION:
Randomized, prospective clinical trial. One group was intervened with povidone-iodine at 5% and the other at 1% as antiseptic for anti-VEGF intravitreal injection. Each patient was evaluated before and after the injection of anti-VEGF for tear break up time, bulbar redness and ocular surface satining with fluorescein. Pain perception was also evaluated 15 minutes after the injection and 48 hours after.

ELIGIBILITY:
Inclusion Criteria

* Having anti-VGEF intravitreal injection scheduled
* Informed consent signed

Exclusion Criteria

* Under 45 years
* Opacity that prevents ophthalmological evaluation and fixation
* Patients with severe dry eye
* Patients with signs of infection on the ocular surface
* Allergy to iodine
* Pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Tear breaking rupture | Change from baseline measured to 15 minutes post-injection
  NIKBUT was measured with Keratopgraph before and after intravitreal injection
Bulbar redness | Change from baseline measured to 15 minutes post-injection
  Bulbar redness was measured with Keratopgraph before and after intravitreal injection

SECONDARY OUTCOMES:
Oxford scale | Change from baseline measured to 15 minutes post-injection
  Oxford scale was measured with fluorescein stain before and after intravitreal injection
Pain analog scale | Change from baseline measured to 15 minutes post-injection
  Pain using visual analog scale was measured 15 minutes and 48 hours after intravitreal injection

CONTACTS AND LOCATIONS:
Overall Officials: José Gerardo García-Aguirre, Principal Investigator — Asociación para Evitar la Ceguera en México I.A.P.
Locations (1):
- Asociación para Evitar la Ceguera en México I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No